CLINICAL TRIAL: NCT04596449
Title: Relationships Between Sleep Spindle and Cognitive Process in Healthy Adults
Acronym: FUSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2020/24
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Sleep
Keywords: Sleep spindles; cognitive processes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Other: study intervention

INTERVENTIONS:
Other: study intervention — The sleep structure of healthy volunteers will be recorded (9 Electroencephalograms (EEG), 2 Electrooculograms (EOG), 2 Electromyograms (EMG) and 2 Electrocardiograms (ECG)) during 1 night. The characteristics of the spindle (density, frequency and amplitude) will be automatically analyzed from purified EEG during Non Rapid Eye Movement sleep (NREM).
  Volunteers will completed a neuropsychological evaluation that will evaluate Sustained attention (simple reaction time test), Vigilance (TAP Vigilance), Sustained and selective attention (CPT II), Inhibition (Stroop test), Mental flexibility (TAP flexibility) , Executive operation (Tower of London), Short-term memory (Wechsler code test).
  Driving performance will be analyzed as part of a complex scenario involving attentional and high-level functions on a driving simulator.

SUMMARY:
Meta-analyses demonstrate that sleep spindles, characterizing NREM sleep, may be a physiological index of high-level cognitive processes. The aim of the study is to determine if sleep spindles can predict interindividual variation in attention and cognitive performance. Relationship between attention and cognitive performance and sleep spindles characteristics (density, frequency and amplitude) recording during 1 night in 80 healthy subject (aged between 18-75y), will be calculated.

DETAILED DESCRIPTION:
It is currently well demonstrated that sleep promotes brain plasticity and therefore is directly involved in cognitive processes such as memory, language, reasoning, learning, intelligence, problem solving…. Sleep deprivation affects most cognitive processes. More specifically, it is the sleep microstructure and in particular the sleep spindles that are specifically linked to memory, learning and cognitive abilities. Sleep spindles are grapho-elements that characterize NREM sleep. They exhibit high inter-individual stability and variability, depend on the genetic heritage and correlate with anatomical properties of the brain. Sleep spindles can therefore be considered as an electrophysiological "finger-print" as one of the most heritable traits of humans. Studies support the notion that sleep spindles are electrophysiological markers of high-level cognitive abilities. It remains to be seen whether the sleep spindles can predict interindividual variations in attention and executive functions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 to 75,
* BMI between 18 and 27,
* Having no subjective daytime sleepiness (Epworth scale score ≤ 11),
* Subjects affiliated to a social security scheme,
* Subjects capable of understanding the study,
* Subjects available to come to the 2 visits required by the study,
* Having given written informed consent to participate in the study,
* Free, informed and written consent, dated and signed by the patient and the investigator before any examination required by the research,
* For simulated driving sub-study: Having a driving license (subsample).

Exclusion Criteria:

* Severe pathologies involving the short-term vital prognosis,
* Uncontrolled endocrine pathologies (dysthyroidism, diabetes),
* All progressive cardiovascular conditions,
* All progressive neurological conditions treated or not (brain tumor, epilepsy, migraine, stroke, sclerosis, myoclonus, chorea, neuropathy, muscular dystrophies, myotonic dystrophy ...),
* Current Psychiatric disorder: mood disorder (depression, bipolar disorder), anxiety disorder, psychosis
* Substance-related dependence,
* Shift workers or night workers who have been on call or on call in the last 72 hours,
* Psychotropic patients,
* Long-term treatment with benzodiazepines and z-drugs,
* Patients on cardiotropic,
* Deprived of liberty by a judicial or administrative decision,
* Pregnant or lactating woman,
* Subject under curatorship or tutorship.
* For simulated driving sub-study: Having simulator-sickness during the first practice session evaluated by Simulator Sickness Questionnaire (SSQ)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Sleep spindle during N2 sleep stage | during experimental visit (between day 1 and day 14 after inclusion)
  Characteristics of the sleep spindles generated during the N2 sleep stages. The sleep spindles density will be calculated automatically on the EEG Cz and Fz channels.
  The amplitude and frequency will be calculated automatically on the EEG Cz and Fz channels.
  The sleep spindles will also be divided, according to their frequency: into fast zones (13-15 Hz) and slow zones (11-13 Hz).
Sleep spindle during N3 sleep stage | during experimental visit (between day 1 and day 14 after inclusion)
  Characteristics of the sleep spindles generated during the N3 sleep stage. The sleep spindles density will be calculated automatically on the EEG Cz and Fz channels.
  The amplitude and frequency will be calculated automatically on the EEG Cz and Fz channels.
  The sleep spindles will also be divided, according to their frequency: into fast zones (13-15 Hz) and slow zones (11-13 Hz).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided